CLINICAL TRIAL: NCT03478670
Title: Adenosine Deaminase Severe Combined Immunodeficiency (ADA-SCID) Registry for Patients Treated With Strimvelis (Previously GSK2696273) Gene Therapy: Long-Term Prospective, Non-Interventional Follow-up of Safety and Effectiveness
Brief Title: Strimvelis Registry Study to Follow-up Patients With Adenosine Deaminase Severe Combined Immunodeficiency (ADA-SCID)
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione Telethon (Other)
Responsible Party: Sponsor
Other Study IDs: STRIM-003
Record Dates: First submitted 2018-03-23; First posted 2018-03-27 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Immunologic Deficiency Syndromes
Keywords: gene therapy; retroviral vector; inherited immune disorder; ADA-SCID; previously GSK2696273; Strimvelis
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Severe combined immunodeficiency due to adenosine deaminase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADA-SCID subjects treated with Strimvelis: Subjects with ADA-SCID who have received Strimvelis (previously GSK2696273) gene therapy, comprising patients treated prior to marketing authorisation (i.e. clinical studies and compassionate use programs) and those treated after marketing authorisation (including within compassionate use and early access programs).
  Interventions: Genetic: Strimvelis

INTERVENTIONS:
Genetic: Strimvelis — Strimvelis is a CD34+ cell enriched dispersion of human autologous bone marrow derived hematopoietic stem/progenitor cells transduced with a retroviral vector containing the human ADA gene. It will be administered as an intravenous infusion once only.
  This is an observational registry that includes all patients who have previously received Strimvelis™ or GSK2696273.

SUMMARY:
Adenosine deaminase (ADA) enzyme deficiency results in severe combined immunodeficiency (SCID), a fatal autosomal recessive inherited immune disorder. Strimvelis (or GSK2696273) is a gene therapy intended for patients with ADA-SCID and for whom no suitable human leukocyte antigen (HLA) matched related stem cell donor is available. This therapy aims to restore ADA function in hematopoietic cell lineages, and in doing so prevents the pathology caused by purine metabolites (i.e., impaired immune function). This registry evaluates the long term safety and effectiveness outcomes of subjects who have received Strimvelis (or GSK2696273).

DETAILED DESCRIPTION:
This is a prospective, non-interventional follow-up registry of patients with ADA-SCID treated with Strimvelis™. The registry does not have a comparator group and the product will have been given on a single occasion prior to entering this registry. Safety and effectiveness will be assessed for a target number of 50 patients who will have received Strimvelis™ (or GSK2696273) comprising patients treated prior to marketing authorisation (i.e. clinical studies and compassionate use programs) and those treated after marketing authorisation (including within compassionate use and early access programs). The registry will close to enrolment when 50 patients have been enrolled but will not close completely until the 50th patient finishes their 15 year follow-up.

ELIGIBILITY:
Inclusion Criteria

1. Patient with ADA-SCID, treated with Strimvelis™ or GSK2696273, as part of its clinical development program.
2. Adult patients, or patients for whom their parents or legal guardians have signed the informed consent form for participation in the registry.

There are no formal exclusion criteria for participation as this registry will follow all patients who have received Strimvelis™ prior to enrollment, subject to informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This registry will include all subjects who have received Strimvelis (or GSK2696273) and consented to participate in the registry. A target number of 50 subjects will be enrolled in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2037-05-31 (Estimated); Study Completion 2037-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | After 15 years of follow-up, it will continue to be solicited every 2 years until the registry closes
  Number and causes of death and time of onset of fatal events will be summarized. Starting time will be the date of therapy administration.
Intervention free survival | Up to 15 years
  Intervention is defined as hematopoietic stem cell transplantation (HSCT) or >3 months of enzyme replacement therapy (ERT)
Number of subjects with the use of medications/treatments of interest | Up to 15 years
  Subjects requiring ERT, HSCT, radiotherapy or cytotoxic agents will be assessed
Absolute peripheral lymphocyte for Immune reconstitution assessment | Up to 15 years
  Peripheral lymphocyte will be assessed
Absolute cluster of differentiation (CD)3+ T-cell for Immune reconstitution assessment | Up to 15 years
  CD3+ T-cell counts will be assessed
Absolute CD19+ B-cell counts for Immune reconstitution assessment | Up to 15 years
  CD19+ B-cell counts will be assessed
Phytohaemagglutinin (PHA) and anti CD-3 as a measure for T cell function | Up to 15 years
  Phytohaemagglutinin (PHA) and anti CD-3 will be assessed
Growth percentile in body height | Up to 15 years
  Subject's height will be superimposed against gender specific World Health Organization (WHO) standard growth charts
Growth percentile in body weight | Up to 15 years
  Subject's weight will be superimposed against gender specific WHO standard growth charts
Deoxyadenosine nucleotides (dAXP) levels in red blood cells for the measurement of systemic metabolite detoxification | Up to 15 years
  Deoxyadenosine nucleotides (dAXP) levels will be assessed in red blood cells
Vector copy number measured in peripheral blood mononuclear cells (PBMCs) | Up to 15 years
  Vector copy number will be measured
Number of subjects with severe infections | Up to 15 years
  Severe infection is defined as an infection requiring hospitalization or prolonging hospitalization
Percentage of subjects with severe infections | Up to 15 years
  Severe infection is defined as an infection requiring hospitalization or prolonging hospitalization
Length of hospital stay | Up to 15 years
  Duration of the hospitalization will be monitored
Number of subjects with non-immunological manifestations of ADA SCID | Up to 15 years
  Subjects will be examined for hepatic steatosis, cognitive deficits, behavioural abnormalities including suspected or diagnosed attention deficit hyperactivity disorder, autism, or hearing impairment
Pediatric development and quality of life data | Up to 15 years
  Determination of attendance at school, if appropriate for age; whether the child is in an age appropriate grade/class at school; whether the child requires special educational support (example [e.g.] dedicated tutor); participation in sports as desired by child; requirement for hearing aid(s); adequate response to childhood vaccinations; severity of impact of a child's health on the guardian's intended employment and Karnofsky/Lansky performance status
Scores for Pediatric Quality of Life Questionnaire (Peds-QL) | Up to 15 years
  Where they are used routinely as part of a physician's standard of care or where permitted by local authorities as non-interventional assessments. The Peds-QL is a generic Health-Related Quality of Life (HR QoL) instrument designed specifically for a pediatric population. It captures the following domains: general health/activities, feelings/emotional, social functioning, school functioning. Higher scores indicate better quality of life (QOL) for all domains of the Peds-QL. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored.
Scores for Ages and Stages Questionnaire-3[ASQ-3] | Up to 15 years
  Where they are used routinely as part of a physician's standard of care or where permitted by local authorities as non-interventional assessments. The ASQ-3 includes a series of questions designed to assess 5 areas of development: communication, gross motor, fine motor, problem solving, and personal social. The questions target behaviours that are appropriate for particular developmental milestones.
Number of subjects with adverse events of interest | Up to 15 years (oncogenesis will continue to be solicited every 2 years until the registry closes)
  AEs and SAEs related to medical or surgical procedures associated with Strimvelis™ administration (e.g. central venous catheter, busulfan conditioning); oncogenesis, autoimmunity, unsuccessful response to gene therapy, hypersensitivity to the product, risks related to residuals present in the drug product administered to the patient, risks related to short shelf-life of product, non-immunologic manifestations of ADA-SCID (e.g. hepatic steatosis, cognitive defects, behavioural abnormalities, hearing impairment), replication competent retrovirus.
Number of subjects with any adverse events (AEs) and any serious adverse events (SAEs) as a safety measure | Up to 15 years
  AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgement will be categorized as SAE
Number of subjects with abnormal clinical laboratory blood test results as a safety measure | Up to 15 years
  Biochemistry, hematology and TSH parameters were assessed
Number of subjects with fertility and pregnancy related outcomes | After 15 years of follow-up, it will continue to be solicited every 2 years until the registry closes
  Labor and delivery information, full term pregnancy, caesarean section, abortion, miscarriage, ectopic, stillbirth rates will be assessed. Both male and female fertility issues will be analyzed.
Data from Retroviral Insertion Site (RIS) analysis and replication competent retrovirus (RCR) | Up to 15 years
  RIS and RCR will be performed when suspected malignancy or after a diagnosis of malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Fondazione Telethon, Study Director — Fondazione Telethon
Locations (1):
- Ospedale San Raffaele, Milan, Lombardy, Italy

REFERENCES:
- [Derived] Migliavacca M, Barzaghi F, Fossati C, Rancoita PMV, Gabaldo M, Dionisio F, Giannelli S, Salerio FA, Ferrua F, Tucci F, Calbi V, Gallo V, Recupero S, Consiglieri G, Pajno R, Sambuco M, Priolo A, Ferri C, Garella V, Monti I, Silvani P, Darin S, Casiraghi M, Corti A, Zancan S, Levi M, Cesana D, Carlucci F, Pituch-Noworolska A, AbdElaziz D, Baumann U, Finocchi A, Cancrini C, Ladogana S, Meinhardt A, Meyts I, Montin D, Notarangelo LD, Porta F, Pasquet M, Speckmann C, Stepensky P, Tommasini A, Rabusin M, Karakas Z, Galicchio M, Leonardi L, Duse M, Guner SN, Di Serio C, Ciceri F, Bernardo ME, Aiuti A, Cicalese MP. Long-term and real-world safety and efficacy of retroviral gene therapy for adenosine deaminase deficiency. Nat Med. 2024 Feb;30(2):488-497. doi: 10.1038/s41591-023-02789-4. Epub 2024 Feb 14. PMID 38355973